CLINICAL TRIAL: NCT00507988
Title: Complex Problem Solving Training in Schizophrenic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Irmtraut Gürkan, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01GW0630
Record Dates: First submitted 2007-07-25; First posted 2007-07-27 (Estimated); Last update posted 2009-05-15 (Estimated); Status verified 2009-05

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Cognitive Training; Complex Problem Solving; Goal Management; Planning
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Complex Problem Solving Training
  Interventions: Behavioral: Complex Problem Solving Training
- B (Active Comparator): Basic Cognitive Training
  Interventions: Behavioral: Basic Cognitive Training

INTERVENTIONS:
Behavioral: Complex Problem Solving Training — 10 sessions of 45 minutes complex problem solving training over 3 weeks (including 30 minutes of computerized planning and problem-solving training with Plan-A-Day and 15 minutes group session for transfer to everyday situations)
  Arms: A
Behavioral: Basic Cognitive Training — 10 sessions over 3 weeks of 45 min basic cognitive training (including 45 min computerized training of attention, processing speed, memory)
  Arms: B

SUMMARY:
The primary purpose of the study is to assess whether a planning and problem-solving training is more effective in improving work therapy performance in patients with schizophrenia than traditional training programs addressing basic cognitive functions.

DETAILED DESCRIPTION:
In patients with schizophrenia, cognitive deficits often lead to an impairment in daily life. This observation has led to the development of cognitive training packages aiming a improving these deficits. However, it is far from clear which level of cognitive functioning provides the best target for cognitive interventions. Traditionally, training has aimed a basic cognitive functions like attention and memory. In the present study we aim at a higher-level of function, namely planning and problem-solving skills, which are trained using the software package Plan-A-Day. The primary hypothesis is that complex problem solving training improved functional capacity more than traditional training programs addressing basic cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Patients with schizophrenic or schizoaffective Disorder (DSM IV)
* Remitted positive symptoms (PANSS positive all ≤ 4), clinical stability
* Native German speaker
* Verbal IQ > 80
* Visual acuity normal or corrected to normal

Exclusion Criteria:

* Concurrent Axis-I disorder
* Drug abuse during last 2 months
* Neurological or medical conditions potentially affecting cognition

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2007-08; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Functional Capacity as assessed by Osnabrücker Arbeitsfähigkeitsprofil "learning ability" subscale | 3 weeks

SECONDARY OUTCOMES:
Functional Capacity as assessed by the Osnabrücker-Arbeitsfähigkeitsprofil summary score | 3 weeks
BADS Zoo Map Score (Neuropsychological Test) | 3 weeks
Planungstest (Tower of London) Summary Score (Neuropsychological Test) | 3 weeks
Plan-A-Day S Solution Time (Neuropsychological Test) | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Weisbrod, MD, Principal Investigator — SRH Klinikum Karlsbad-Langensteinbach, Department of Psychiatry
Locations (1):
- SRH Klinikum Karlsbad-Langensteinbach, Karlsbad, Germany

REFERENCES:
- [Derived] Rodewald K, Rentrop M, Holt DV, Roesch-Ely D, Backenstrass M, Funke J, Weisbrod M, Kaiser S. Planning and problem-solving training for patients with schizophrenia: a randomized controlled trial. BMC Psychiatry. 2011 Apr 28;11:73. doi: 10.1186/1471-244X-11-73. PMID 21527028